CLINICAL TRIAL: NCT04128670
Title: Effects of Kinesio Tape on Delayed Onset Muscle Soreness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kelly Naugle, PhD, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1908530527
Record Dates: First submitted 2019-10-11; First posted 2019-10-16 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Delayed Onset Muscle Soreness
Keywords: kinesio tape; muscle soreness; eccentric exercise; muscle pain
MeSH Terms: conditions — Myalgia | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Randomized single-blind controlled trial
Who Masked: Participant
Masking Description: Participant will not know if they are in the experimental taping condition or the placebo taping condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Kinesiotape (KT) (Experimental): Tape will be applied to the biceps muscle of the nondominant arm from approximately the shoulder to the elbow for up to 72 hours. For the KT group taping will be applied with a lymphatic application method according to the guidelines recommended by Kenzo Kase. This type of application is known to improve blood and lymphatic circulation which enhances the removal of metabolic products. The tape will be applied with a tension of 10-20%.
  Interventions: Device: Kinesiotape
- Placebo Kinesiotape (Placebo Comparator): Tape will be applied to the biceps muscle of the nondominant arm from approximately the shoulder to the elbow for up to 72 hours. The placebo KT group will have 0% tension.
  Interventions: Device: Kinesiotape
- No Tape (No Intervention): This group will not receive any intervention.

INTERVENTIONS:
Device: Kinesiotape — Tape will be applied to the biceps muscle of the nondominant arm from approximately the shoulder to the elbow for up to 72 hours. For the KT group taping will be applied with a lymphatic application method according to the guidelines recommended by Kenzo Kase. This type of application is known to improve blood and lymphatic circulation which enhances the removal of metabolic products. It is recommended that the application of the tape for lymphatic correction be applied for 24-72 hours. The tape will be applied with a tension of 10-20%.
  Arms: Kinesiotape (KT); Placebo Kinesiotape

SUMMARY:
The purpose of this study is to determine the effect of Kinesio tape on delayed onset muscle soreness of the biceps muscle of your arm following strenuous exercise of the bicep muscle.

DETAILED DESCRIPTION:
Participants will complete 4 testing sessions that will be held on 4 separate days (Baseline, Eccentric Exercise day, 48 hours post exercise, and 72 hours post exercise). All sessions will take place in the National Institute of Fitness and Sport, where the Department of Kinesiology laboratories are located.

During the first session (Baseline), the purpose and procedures of the research will be explained by the investigator, co-investigator, or a research assistant in more detail. Participants will read and sign the informed consent form and then undergo an exclusion/inclusion criteria assessment which includes the Physical Activity Readiness Questionnaire (PAR-Q), and brief questionnaire. All study personnel/staff obtaining informed consent will be trained in the responsible conduct of research. All participants will be asked if they have a known allergy to Kinesio Tape (KT) or if they have sensitive skin. Those with sensitive skin will be administered an allergy test. After screening and enrollment, participants will complete baseline assessments of muscle pain and function, pain sensitivity, and psychological risk factors (See outcome measures).

During Session 2, strength of the non-dominant bicep will be measured first. Participants will then perform an eccentric exercise protocol designed to induce delayed onset muscle soreness (DOMS) on the non-dominant arm. Strength of the non-dominant bicep will be measured immediately post the eccentric exercise protocol. At the end of this session, subjects will be randomly assigned to one of two intervention groups (experimental KT group, placebo KT group) or a control group (i.e., no intervention performed). The experimental group will receive KT with proper technique and tension (10-20%), while the placebo group will receive KT without technique and tension.

Sessions 3 and 4 will occur approximately 48 and 72 hours post Session 2, respectively. All the outcome variables will be measured during these sessions. For participants in the KT groups, the tape will be removed at the end of session 4, as described below.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30 years old

Exclusion Criteria:

* Participating in any strengthening exercises or activities of the upper extremities for the past month.
* Regularly (~2x per month) participating in strengthening exercises or activities that include lengthening actions of the upper extremity for the past 6 months.
* An answer of yes to any of the seven questions on the first page of the 2019 Physical Activity Readiness Questionnaire [PAR-Q: 16] indicating that the subject is not physically ready for exercise without a medical exam. These exclusions include the following:

  * If participant's doctor has ever said that he/she has a heart condition or high blood pressure
  * Pain in chest at rest, during daily activities of living, or when doing physical activity
  * If participant has ever lost balance because of dizziness or has lost consciousness in the past 12 months
  * If the participant currently has (or have had within the past 12 months) a bone, joint, or soft tissue (muscle, ligament, or tendon) problem that could be made worse by becoming more physically activity
  * If participant is currently taking prescribed medications for a chronic medical condition
  * If the participant's doctor has ever told them that they should only do medically supervised physical activity.
* Currently taking nutritional supplements or anti-inflammatory medication on a daily basis
* Any injury or surgery to the neck or upper extremity in the past 6 months
* Open or scabbed wounds in the arm area to be taped
* Known allergies to the tape or medical adhesive bandages
* If skin irritation develops to the tape

Session exclusion criteria:

● Taking over-the-counter pain medications on days of testing, prior to testing sessions, including acetaminophen (Tylenol) and nonsteroidal inflammatory drugs (NSAIDs), including ibuprofen (Motrin, Advil) or naproxen (Aleve, Naprosyn).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
change in worst pain in previous 24 hours | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  Brief Pain Inventory
Change in average pain in previous 24 hours | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  Brief Pain Inventory
Change in pain during elbow extension and elbow flexion | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  Subjects will perform the following elbow movements: 1) moving from a fully flexed starting position through active range of motion to full extension 2) moving from a fully extended starting position through active range of motion to full flexion. Ratings of muscle pain intensity will be assessed following each contraction using a 0-100 scale, with "0" indicating "no pain" and "100" indicating the "most intense pain imaginable".
Change in pressure pain threshold of the affected biceps | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  Using a hand-held, clinical grade pressure algometer (Wagner Instruments, Greenwich, CT), pressure will be applied to the biceps brachii muscle of the affected (non-dominant) arm while the arm is stationary at approximately 90 degrees of elbow flexion. Pressure will increase at a rate of about 1kg/s until the subject first reports feeling pain.
Change in Active Total Elbow Range of Motion (AT-ROM) | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  AT-ROM in elbow flexion and extension of the elbow joint will be measured with a standard goniometer and the subject in the supine position on a padded table. The subject is instructed to flex and extend the non-dominant arm at the elbow "as far as you can". Elbow flexion and extension is assessed in the sagittal plane with the arm parallel to the trunk and in the anatomic position. The center fulcrum of the goniometer is placed over the lateral epicondyle of the humerus. The stationary arm of the goniometer is fixed along the lateral midline of the humerus in line with the acromion process and the moving arm along the lateral midline of the radius in the line with the styloid. Three measurements of active elbow flexion and extension will be conducted at each assessment time point, with the average of the three measurements used as the outcome measure for each time point.
Change in pain during elbow flexion and extension | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  Subjects will perform the following elbow movements: 1) moving from a fully flexed starting position through active range of motion to full extension 2) moving from a fully extended starting position through active range of motion to full flexion. Ratings of muscle pain intensity will be assessed following each contraction using a 0-100 scale, with "0" indicating "no pain" and "100" indicating the "most intense pain imaginable".
Change in Maximal Strength of non-dominant bicep. | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  Maximal strength will be assessed by performing a maximal contraction with the arm flexed at 90 degrees. The participant will be seated on a Biodex strength testing machine, with both feet on a support and the upper arm supported at 45 degrees of shoulder flexion by a padded support arm, with the forearm flexed at 90 degrees during the contraction. Three maximal contractions will be performed at 60 degrees per second with 60 seconds of rest between trials.

SECONDARY OUTCOMES:
Change in Self-reported function of the affected arm | This measure will be assessed at baseline and 48 hours and 72 hours following completion of the eccentric exercise protocol
  The QuickDASH focuses on the subject's ability to use the affected arm during activities of daily living [23,24]. Subjects rate their symptoms and ability to perform specific tasks using a 5-pt hierarchical Likert scale. A score of zero represents no dysfunction at all, while higher scores represent more limitations in self-reported function, with a score of 100 being the highest possible score.
Pain catastrophizing | This instrument will be administered at baseline
  Will be measured with the Pain Catastrophizing Scale. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Fear of movement or reinjury | This instrument will be administered at baseline
  Will be measured with the Tampa Scale of Kinesiophobia -- (TSK-11). total TSK-11 scores range from 11-44 points with higher scores indicating greater fear of pain, movement, and injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Purdue University Indianapolis, Indianapolis, Indiana, United States